CLINICAL TRIAL: NCT01350284
Title: Effect of Cinnamon on Gastric Emptying, Arterial Stiffness, Postprandial Lipaemia, Glycaemia, and Appetite Responses to High-fat Breakfast
Brief Title: The Effect of Natural Food Flavourings on Gastrointestinal and Cardiovascular Physiological Responses.
Acronym: CinnGastEmpt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: University of Ulster (Other); Ulster Hospital, Northern Ireland (Unknown); National University of Ireland, Galway, Ireland (Other)
Responsible Party: Amir Shafat, PhD, University of Limerick
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CinnGastEmpt
Record Dates: First submitted 2011-05-03; First posted 2011-05-09 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-05

CONDITIONS: Gastric Emptying; Diabetes Mellitus
Keywords: Antioxidants; Glucose Intolerance prevention and control; Diabetes Mellitus prevention and control
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dietary supplementation (Experimental): 3g of cinnamon or placebo control were added to a test-meal.
  Interventions: Dietary Supplement: Cinnamon; Dietary Supplement: Placebo control

INTERVENTIONS:
Dietary Supplement: Cinnamon — acute oral administration of 3 g cinnamon
Dietary Supplement: Placebo control — 3 g wheat flour (placebo)- separated by 28 days from cinnamon intervention

SUMMARY:
The purpose of this study is to determine whether 3 g cinnamon was sufficient to delay the gastric emptying rate of a high-fat solid meal and subsequently reduce postprandial blood glucose and lipid responses, oxidative stress, arterial stiffness and satiety responses in a healthy adult population.

DETAILED DESCRIPTION:
Cinnamon has been shown to delay gastric emptying (GE) of a high-carbohydrate meal and reduce postprandial glycaemia in healthy adults. However, it is dietary fat which is implicated in the etiology and is associated with obesity, type 2 diabetes (T2D) and cardiovascular disease (CVD). We aimed to determine the effect of 3 g cinnamon on GE, postprandial lipemic and glycemic responses, oxidative stress, arterial stiffness, as well as appetite sensations and subsequent food intake following a high-fat (HF) meal.

The effect of acute oral administration of 3 g cinnamon on gastric emptying of a high-fat pancake test meal and subjective appetite sensations by visual analogue scale will be measured for six hours postprandially. During this time course, measurements of postprandial lipemic, glycemic, oxidative stress and arterial stiffness responses will be collected. Subsequently, food intake will be measured using an ad libitum buffet meal. The study will be conducted in a randomized, placebo-controlled, single-blinded manner in 9 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-35 years
* Recreationally trained individuals (participate in at least 2hrs/wk of individual/team sport)
* Not currently taking antioxidant or lipid-lowering medication
* Fasting blood lipid, glucose and blood pressure (BP) levels were all within the normal limits.

Exclusion Criteria:

* History of gastrointestinal-related conditions, diabetes mellitus or cardiovascular disease.
* Allergies to foods in study.
* Blood disorder
* Pregnancy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The effect of 3grams cinnamon on gastric emptying half time | During the 6.5 hours post ingestion

SECONDARY OUTCOMES:
Arterial stiffness | During the 6.5 hours after ingestion
  Post-prandial changes in pulse wave velocity (m/s) will be measured non-invasively, using Pulsetrace PSA2 to indicate arterial stiffness.
Lipaemia | During the 6.5 hours after ingestion
  Plasma concentration (mmol/l) of triacylglycerols, LDL, and HDL will be measured every hour in the post-prandial period.
Glycemia | During the 6.5 hours after ingestion
  The concentration of plasma glucose (mmol/l) will measured hourly in the postprandial period, using venous blood drawn from a forearm vein.
Appetite | During the 6.5 hours after ingestion
  Subjective sensation of hunger, desire to eat, fullness, thirst, tiredness and coldness will be meaured using a 150mm visual analogue scale (mm).
Oxidative stress | During the 6.5 hours after ingestion
  Serum lipidhydroperoxides will be measured using FOX-1 assay.
Food intake | 6 hours post-prandially
  A buffet meal will be presented to the volunteer 6h after breakfast. Food intake will be monitored covertly by weighing individiual food items before and after presentation. Food intake will be expressed as macronutrient (carbohydrate, fat, protein, water, fibre) and energy intake.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Shafat, PhD, Principal Investigator — Univeristy of Limerick
Locations (1):
- Department of Physical Education & Sport Sciences, University of Limerick, Limerick, Ireland

REFERENCES:
- [Derived] Markey O, McClean CM, Medlow P, Davison GW, Trinick TR, Duly E, Shafat A. Effect of cinnamon on gastric emptying, arterial stiffness, postprandial lipemia, glycemia, and appetite responses to high-fat breakfast. Cardiovasc Diabetol. 2011 Sep 7;10:78. doi: 10.1186/1475-2840-10-78. PMID 21899741